CLINICAL TRIAL: NCT05397860
Title: Radiofrequency Ablation for Hepatocellular Carcinoma Using Gradual Radiofrequency (RF) Energy Delivery Mode With Octopus Electrodes: A Prospective Observational Study
Brief Title: Radiofrequency Ablation With Gradual Radiofrequency Energy Increment for Hepatocellular Carcinoma Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Starmed (Industry)
Responsible Party: Principal Investigator, Jeong Min Lee, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1909-086-1064
Record Dates: First submitted 2022-05-26; First posted 2022-05-31 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Hepatocellular Carcinoma; Liver Cirrhosis; Chronic Liver Disease
Keywords: Radiofrequency ablation; Gradual radiofrequency energy increment; Cone-unit ablation
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Cirrhosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with clinically diagnosed hepatocellular carcinoma (HCC) (equal or less than 4 cm ) (Experimental): Patients with chronic hepatitis B or liver cirrhosis have hepatocellular carcinoma (HCC) (equal or less than 4 cm) which is diagnosed on contrast-enhanced computed tomography (CT) or magnetic resonance imaging (MRI).
  Interventions: Procedure: Radiofrequency ablation using gradual radiofrequency energy delivery with Octopus electrodes

INTERVENTIONS:
Procedure: Radiofrequency ablation using gradual radiofrequency energy delivery with Octopus electrodes — Radiofrequency ablation (RFA) will be performed by using multi-VIVA generator and Octopus electrodes. Three electrodes will be placed on the tumor under ultrasonography (US)-computed tomography (CT)/magnetic resonance (MR) fusion tool guidance. The electrodes will be cooled with saline, and radiofrequency (RF) will be applied to two of three electrodes at the same time for about 6 to 30 minutes depending on the tumor size. The temperature will be maintained at 90-100 °C. The RF energy will starts at 60 watts and increase by 10 watts every 30 seconds for the first 3 minutes, and then increases gradually by 10 watts per minute after reaching 100 watts.

SUMMARY:
To evaluate local tumor progression rate at 12 months after percutaneous radiofrequency ablation with gradual radiofrequency energy delivery mode with Octopus electrodes in patients with hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Child-Pugh Class A or B
* chronic hepatitis B or liver cirrhosis
* contrast enhanced computed tomography (CT) or magnetic resonance imaging (MRI) within 60 days of scheduled radiofrequency ablation (RFA) date
* clinically diagnosed hepatocellular carcinoma (HCC), equal or less than 4 cm

Exclusion Criteria:

* number of HCC, equal or more than 3
* largest tumor size over 4 cm
* Child-Pugh class C
* presence of vascular invasion by HCC
* platelet count less than 40,000 per mm3 or International Normalized Ratio (INR) prolongation over 50%
* presence of extrahepatic metastasis

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-01-06 (Actual); Primary Completion 2023-08-30 (Estimated); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
Local tumor progression rate | 12 months after radiofrequency ablation (RFA)
  Evaluate local tumor progression by follow-up computed tomography (CT) or magnetic resonance imaging (MRI) with alpha-fetoprotein (AFP) level

SECONDARY OUTCOMES:
Success rate of cone-unit ablation | Immediately after radiofrequency ablation (RFA)
  The cone-unit ablation is defined as complete ablation of tumor with safety margin and occlusion of the 4th or 5th branches of portal vein.

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Min Lee, M.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hwang S, Kim JH, Yu SJ, Lee JM. Incremental high power radiofrequency ablation with multi-electrodes for small hepatocellular carcinoma: a prospective study. BMC Gastroenterol. 2024 Aug 21;24(1):280. doi: 10.1186/s12876-024-03358-w. PMID 39169297
- [Derived] Kim JH, Kim HS, Yoon JH, Joo I, Yoon JH, Kim YJ, Yu SJ, Lee JM. Anatomical ablation for small hepatocellular carcinomas using multiple applicators: a preliminary study. Cancer Imaging. 2023 Aug 21;23(1):78. doi: 10.1186/s40644-023-00597-0. PMID 37605251